CLINICAL TRIAL: NCT05319249
Title: Natural Killer Cell Immunotherapy in Combination With PARP-inhibition to Overcome NKG2D Mediated Immune Evasion in Acute Myeloid Leukemia
Brief Title: Natural Killer Cell Immunotherapy in Combination With PARP-inhibition in Acute Myeloid Leukemia
Acronym: NAKIP-AML
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAKIP_01_2022
Record Dates: First submitted 2022-03-21; First posted 2022-04-08 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — talazoparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NK cells combined with PARP inhibition (Experimental): Combination of NK cell therapy and PARP inhibition by Talazoparib after immunosuppression with cyclophosphamide and fludarabine
  Interventions: Biological: NK cells; Drug: Talazoparib 1 MG [Talzenna]

INTERVENTIONS:
Biological: NK cells — NK cells will be given as a single intravenous infusion.
  Other Names: Haploidentical human allogeneic NK cells
Drug: Talazoparib 1 MG [Talzenna] — Subjects will receive treatment with Talazoparib capsules 1 mg/day (4 days) with subsequent intravenous NK cell infusion.
  Other Names: Talzenna

SUMMARY:
Therapy resistance remains the major obstacle to cure in many types of cancer. In particular in leukemia, therapy resistance depends on leukemic stem cells (LSC) that exhibit inherent therapy resistance to multiple drugs and contribute to overt leukemic relapse. Cellular therapies alone or in combination with other targeted or chemotherapeutic approaches can overcome drug mediated therapy resistance and induce long lasting remissions. Several trials have shown that adoptive transfer of allogeneic NK cells can induce clinical remission in patients with myeloid malignancies. In addition, the antileukemic efficacy of alloreactive NK cells has been shown to facilitate cure after T cell depleted haploidentical stem cell transplantation. Recently, it was demonstrated that absence of NKGD2 ligand expression on leukemic stem cells determines therapy resistance and immune escape towards NK cells in AML. PARP1 inhibitors can induce re-expression of NKG2D ligands. This phase I/II clinical trial will evaluate the combination of NK cell therapy and PARP inhibition by Talazoparib in patients with poor prognosis AML as characterized by Minimal Residual Disease (MRD) or overt relapse with less than 20% bone marrow blasts. The hypothesis that allogeneic NK cell therapy combined with PARP inhibition will increase the response rate (CR/CRi for relapsed/ refractory patients and MRD-response for MRD positive patients) from 35% to 60% will be tested. The co-primary endpoints are i) response to treatment defined as complete remission (CR) for patients with overt leukemia at time of inclusion and MRD decrease >1log10 for patients with rising MRD at time of inclusion as well as ii) safety and feasibility of the protocol. Key secondary endpoints are event free survival and overall survival. Two cohorts will be assessed independently: patients with i) overt leukemia and ii) patients with rising MRD at time of inclusion. Safety and feasibility will be analyzed continuously during the entire trial. The NAKIP-AML trial will analyze efficacy and feasibility of NK cell transplantation together with PARP1 inhibition.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed diagnosis of AML according to WHO-2016 (Arber, Orazi et al. 2016) (except acute promyelocytic leukemia) with either de novo AML, AML after preceding myelodysplastic or myeloproliferative syndrome (MDS/MPD), and therapy- related AML (t-AML) after previous cytotoxic therapy or radiation are eligible.

   A) Relapsed or Refractory AML with less than 20% bone marrow blasts and less than 20% blasts in peripheral blood.

   B) Rising MRD levels (>3 fold) as detected by either molecular genetics or flow cytometry in patients still in hematologic remission.
2. Patients who received at least one line of AML therapy. This is defined as either stem cell transplantation or intensive AML therapy or palliative AML therapy containing at least one of the following drugs Azacitidine, Decitabine, Cytarabine, Venetoclax or an FLT3 inhibitor..
3. Discontinuation of prior AML treatment before the start of study treatment for at least 107 days for cytotoxic agents and ≥ 53 half-lives for non-cytotoxic / investigational drug treatment preceding the first dose of trial medications.
4. Age ≥ 18 years
5. ECOG ≤2
6. Pregnancy and childbearing potential:

   * Non-pregnant and non-nursing women of childbearing potential must have a negative serum or urine ß-HCG pregnancy test within a sensitivity of at least 25 mIU/mL within 72 hours prior to registration. ("Women of childbearing potential" is defined as a sexually active mature woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 consecutive months).
   * Female patients of reproductive age must agree to avoid getting pregnant while on therapy.
   * Women of child-bearing potential must either commit to continued abstinence from heterosexual intercourse or begin highly effective methods (referring to recommendation of the CTFG) of birth control during study and at least 6 months (women), after end of treatment.
   * Men must use a latex condom during any sexual contact with women of childbearing potential, even if they have undergone a successful vasectomy and must agree to avoid to father a child during study and until 6 months after end of treatment.
7. Willingness of patients to adhere to protocol specific requirements and capacity to give written informed consent
8. Ability of patient to understand the character and individual consequences of clinical trial
9. Following receipt of verbal and written information about the study, the patient must provide signed informed consent before any study related activity is carried out.
10. Suitable donor for NK cell transplantation

Exclusion Criteria:

Patients presenting with any of the following criteria will not be included in the trial:

1. Acute promyelocytic leukemia (AML M3)
2. AML in which less than 10% of the blasts express the CD34 surface marker expression as analyzed at the local laboratory.
3. Known central nervous system manifestation of AML
4. Uncontrolled or significant cardiovascular disease, including any of the following:

   * Heart failure NYHA class 3 or 4
   * Left ventricular ejection fraction (LVEF) ≤ 40% by echocardiogram ECHO)
   * History of uncontrolled angina pectoris or myocardial infarction within 12 months prior to screening
   * History of second (Mobitz II) or third-degree heart block or any cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
5. Pregnant or nursing women
6. Chronically impaired renal function (creatinine clearance < 30 ml / min)
7. Organ dysfunction (e.g. liver, kidney, lung, heart) which in the opinion of the treating physician decreases life expectancy to less than three months.
8. Kidney failure with a calculated glomerular filtration rate <30 ml/min or bilirubin >2-fold the upper reference limit of the local laboratory.
9. HIV infection and/or active hepatitis B or C infection (active hepatitis B defined by HBs Ag positivity, anti HBs positivity or anti-HBC positivity, active hepatitis C defined by positive virus load).
10. Evidence or history of severe non-leukemia associated bleeding diathesis or coagulopathy
11. Uncontrolled active infection
12. Concurrent malignancies other than AML with an estimated life expectancy of less than two years
13. Known hypersensitivity to PARP inhibitors
14. Isolated extramedullary manifestation of AML
15. Patients < 100 days after allogeneic stem cell transplantation at the time of screening
16. Expected non-compliance of patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
complete remission (CR/CRi) | Collected at a minimum at baseline, day 28 and latest on day 42
  response defined as complete remission (CR/CRi) for patients with overt leukemia at time of inclusion and MRD decrease >1log10 for patients with rising MRD at time of inclusion.

SECONDARY OUTCOMES:
EFS - Event-free survival | EFS is defined as the time of entry into the study to the date of primary refractory disease, or relapse from CR, or CRi, or death from any cause, whichever comes first, assessed up to 42 days.
  Event-free survival
RFS -Relapse-free survival | Defined as the time from achieving a remission until the date of relapse or death from any cause, whichever comes first, assessed up to 42 days.
  RFS is defined only for patients achieving CR or CRi
OS - Overall survival | OS is defined as the time from entry into the trial to the date of death from any cause, assessed up to 42 days.
  Overall survival
MRD | Collected at a minimum at baseline, day 28 and latest on day 42
  Measurable Residual Disease
QoL - Quality of life - QLQ-C30 | QoL is assessed at baseline and latest on day 42.
  Validated 30-item self-assessment questionnaire to assess quality of life aspects. The items are rated on a 4-point Likert scale ranging from 1 (not at all) to 4 (very much) with higher scores meaning a higher level of fatigue.